CLINICAL TRIAL: NCT05250583
Title: Use of a Double Amniotic Membrane Inserted in a Ring of Umbilical Vessels with Wharton's Jelly, Tissues Treated by the AMTRIX Process, in the Treatment of Keratitis Resisting Healing Medical Treatment
Brief Title: Use of a Biological Lens of Amniotic Membrane (LV-Visio-AMTRIX) in the Treatment of Treatment-Resistant Keratitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-Visio-AMTRIX-TBF3; 2019-A03144-53 (Other: IDRCB)
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Keratitis
MeSH Terms: conditions — Keratitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LV-Visio-AMTRIX (Experimental): Sutureless amniotic membrane supported by a biological ring.
  Interventions: Biological: LV-Visio-AMTRIX

INTERVENTIONS:
Biological: LV-Visio-AMTRIX — Chemically-treated, viro-inactivated, freeze-dried and irradiated allograft placed by the investigator during patients' hospital visit

SUMMARY:
The purpose of this open, mono center trial is to assess the impact of the use of an amniotic membrane on the healing of a keratitis resistant to medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; age between 18 and 65 years.
* Patient with non-infectious keratitis resistant to medical treatment for more than 15 days or recurrent after healing treatment.
* Patient with quantitative and qualitative score for inflammatory ocular signs > 20.
* Patient with Oxford grade > 2.
* Informed and consenting patient with a relative or friend available to instill eye drops if necessary.
* Patient affiliated to a social security system or beneficiary of such a system.

Exclusion Criteria:

* Patient with active infectious keratitis (bacterial, parasitic or viral).
* Patient with allergy to Oxybuprocaine or Tetracaine eye drops, to ester type local anesthetics and to fluorescein.
* Current contact lens wear, including scleral lenses.
* NSAID eye drops and any drops containing preservatives.
* Antibiotic, anti-viral, anti-parasitic eye drops.
* Patient with identified causes for the keratitis for which discontinuation of medical treatment beneficial.
* Ocular surgery in the 3 months preceding the inclusion in the study.
* Monophtalmic patient.
* Person deprived of liberty by a judicial or administrative decision.
* Adult subjected to a legal protection measure or unable to express his/her consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Keratitis healing within 15 days after the beginning of the treatment | 15 days
  Keratitis observed under slit lamp using fluorescein instillation. Keratitis considered healed if epithelialization of more than 50% and/or Oxford < grade 2

SECONDARY OUTCOMES:
Stable or decreased score for inflammatory and clinical signs of the ocular surface | 1 day, 3 days, 5 days, 7 days, 10 days, 15 days, 30 days, 45 days
  Composite score for inflammatory and clinical signs of the ocular surface on 66 points. Duration and intensity are evaluated for secretion, dry eyes, tearing, foreign body sensation, fluctuating vision, photophobia, burning sensation and lids edema. Duration is evaluated from a scale from 0: never to 4: all the time. Intensity is evaluated from a scale from 0: slight to 2: severe. Localization and intensity are evaluated for conjunctival edema, conjunctival redness and neovascularization. Localization is evaluated on a scale from 0: no reaction to 4: reaction present in the whole eye.
Stabilisation or decrease of pain evaluated on visual analog scale | 1 day, 3 days, 5 days, 7 days, 10 days, 15 days, 30 days, 45 days
  Visual Analog Scale (VAS) on 10 points from 0: no pain to 10: worst imaginable pain
Preservation of epithelialization | 15 days, 30 days, 45 days
  Preservation of new epithelialization evaluated under slit lamp using fluorescein instillation and Oxford grading system
Change in eye dryness | 15 days, 30 days, 45 days
  Eye dryness evaluated by the Ocular Surface Disease Index (OSDI) (0-12 = normal; 13-22 = mild dry eye; 23-32 = moderate dry eye; >33 = severe dry eye)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Saint-Etienne Hôpital Nord, Saint-Priest-en-Jarez, France